CLINICAL TRIAL: NCT05783245
Title: Effect of Cooling Therapy for Post-Operative Pain in Open Carpal Tunnel Release
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB21-1298
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Carpal Tunnel Syndrome; Perioperative/Postoperative Complications
MeSH Terms: conditions — Carpal Tunnel Syndrome; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Ice Therapy (Experimental): Postoperative care with experimental ice therapy
  Interventions: Other: Polarcare Machine
- Standard of Care Ice Therapy (Active Comparator): Postoperative care with standard of care ice therapy
  Interventions: Other: Standard of care ice therapy

INTERVENTIONS:
Other: Polarcare Machine — Use of Polar Care ice machine as often as possible, but a minimum of three 15 minute uses per day, for the first 3 days after surgery. No single use should last longer than 30 minutes.
  Arms: Experimental Ice Therapy
Other: Standard of care ice therapy — Use of commercial reusable ice packs as often as possible, but a minimum of three 15 minute uses per day, for the first 3 days after surgery. No single use should last longer than 30 minutes.
  Arms: Standard of Care Ice Therapy

SUMMARY:
This study seeks to perform an appropriately-powered study to evaluate any clinical difference between continuous cooling therapy and traditional ice for treatment of post-operative pain in open CTR surgery.

DETAILED DESCRIPTION:
Post-operative pain control is paramount to all operative procedures and involves several modalities. Both pharmaceutical and non-pharmaceutical measures are frequently used. Carpal tunnel release (CTR) surgery is one of the most common surgeries performed in the U.S. with over 400,000 procedures per year.2 Frequently, ice is used as a treatment modality following surgical CTR.3 Several products have been developed in the past decades to improve ice therapy in the rehabilitation period. One such product is the Polar Care which provides up to 6-8 hours of continuous icing.

While there is good data supporting the use of cooling therapy (ice) for post-operative pain, there is lack of data surrounding the use of continuous cooling therapy machines such as the PolarCare following carpal tunnel release (CTR). The two papers that evaluated the efficacy of continuous cooling therapy following CTR had conflicting results on any added benefit of continuous cooling therapy over traditional icing.

There is no standard of care for post-operative icing at UCMC following CTR. Clinicians currently decide whether to give patients a PolarCare machine on the day of surgery without any algorithm. All other patients are encouraged to use traditional icing methods. This study seeks to perform an appropriately-powered study to evaluate any clinical difference between continuous cooling therapy and traditional ice for treatment of post-operative pain in open CTR surgery.

The investigators hypothesize that participants receiving continuous cooling therapy will have a statistically significantly lower pain score compared to those receiving traditional ice therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Indicated for open carpal tunnel release
3. Able and willing to complete online questionnaires

Exclusion Criteria:

1. Prior carpal tunnel surgery for ipsilateral extremity
2. Additional procedures to be performed on ipsilateral or contralateral extremity
3. Current opioid or narcotic pain medication usage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) for pain | 3 days
  The visual analog scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable. A patient marks a point on the line that matches the amount of pain he or she feels.

SECONDARY OUTCOMES:
Disabilities of the Arm, Shoulder, and Hand questionnaire | 1 week
  he DASH is a 30-item self-report questionnaire designed to assess musculoskeletal disorders of the upper limbs.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Wolf, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers